CLINICAL TRIAL: NCT04888325
Title: Effects of Oral vs Intravenous Glucose Administration on Novel Candidates of Energy Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Alexandros Kokkinos, Associate Professor in Internal Medicine, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 284/02-03-2018
Record Dates: First submitted 2021-05-09; First posted 2021-05-17 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Glucose; Glucose Tolerance Test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral glucose (Experimental): ORal glucose consumption 1.25 grams/kg in 200 ml water at time 0 and the same amount again at 3 hours
  Interventions: Other: Oral glucose
- Intravenous glucose (Experimental): 0% intravenous glucose infusion at a rate of 3.6 ml/kg/h
  Interventions: Other: Intravenous glucose

INTERVENTIONS:
Other: Oral glucose — Oral glucose consumption (1.25 grams/kg in 200 ml water at time 0 and the same amount again at 3 hours). During the 6-hour observation period infusion of normal saline (NaCL 0,9%) at a rate of 0.83 plus Heparin, 800 IU/h with a priming dose of 1000 IU.
  Arms: Oral glucose
Other: Intravenous glucose — 10% intravenous glucose infusion at a rate of 3.6 ml/kg/h plus Heparin 800 IU/h with a priming dose of 1000 IU will be administrated for 6 hours. Consumption of 300 ml of water at 0 and 3 hours
  Arms: Intravenous glucose

SUMMARY:
Energy regulation in humans is controlled through complicated mechanisms involving among others hormones secreted from different tissues, such as gut, muscle and adipose tissue. Specifically, the hormonal secretion after nutrient intake mediates the metabolic response in order to maintain energy balance. Proglucagon-derived hormones and especially GLP-1 and glucagon are significantly affected by nutrient intake and by energy balance. Despite the extensive information about GLP-1 and glucagon, it remains unclear whether other proglucagon-derived hormones are regulated by nutrition or by energy status i.e. obesity or type 2 diabetes. Similarly, secretion of activins and follistatins, which are both affecting muscle metabolism-growth and consequently energy homeostasis, are reduced in energy deprivation states. However, we do not know whether the circulating profile of these hormones is affected acutely by nutrient intake and whether these changes have acute effects on muscle metabolism.

We propose to conduct a non-blinded interventional study evaluating the effects of oral or intravenous glucose intake in the circulating levels of proglucagon-derived hormones, activin A, activin B, follistatin, follistatin-like 3.

DETAILED DESCRIPTION:
Screening Visit: Potential subjects will present for a study screening visit in the study site. A written informed consent will be obtained by a study physician at the screening visit. Potential subjects will have their medical history obtained and will be examined by a study physician. Vitals will be taken and height, weight, and waist circumference will be measured. Potential subjects will have a screening fingerstick glucose test as a marker of diabetes and blood collected for CBC and basic lipid panel. Menstrual status will be assessed by menstrual history (female subjects only) and women will take a urine pregnancy test and will be excluded from participation if pregnant. Subjects will meet with a registered dietitian.

Visit 1: Subjects will return to the GCRC after a 10-hour overnight fast. In the study site, subjects will have vital signs and anthropometrics measured. All subjects will have one IV line, used to obtain blood samples for insulin, glucose, proglucagon derived hormones and muscle-acting hormones (activin A, activin B, follistatin, follistatin-like 3).

Participants will consume orally glucose 1.25 grams/kg in 200 ml water at time 0 and the same amount again at 3 hours. During the 6-hour period they are also going to receive normal saline (NaCL 0,9%) at a rate of 0.83 plus Heparin, 800 IU/h with a priming dose of 1000 IU.

Blood collection will be obtained from the IV line at 30 min intervals for the first 2 hrs and hourly thereafter.

Visit 2: Subjects will return after a 10-hour overnight visit. Visit 2 will be performed at least 1 week after Visit 1. All subjects will have two IV lines, one for obtaining blood samples for insulin, glucose, proglucagon derived hormones and muscle-acting hormones (activin A, activin B, follistatin, follistatin-like 3) and another one for the intravenous administration of glucose.

Specifically a 10% intravenous glucose infusion at a rate of 3.6 ml/kg/h plus Heparin 800 IU/h with a priming dose of 1000 IU will be administrated for 6 hours. At time 0 and at 3 hours they will drink 300 ml water to control for any effects of gastric distension.

Blood collection will be obtained from the IV line at 30 min intervals for the first 2 hrs and hourly thereafter.

Each blood draw will be 15 ml (5 ml in EDTA tubes with aprotinin and 10 ml in serum tubes).

ELIGIBILITY:
Inclusion Criteria:

Adult (18-65 years of age) men and women

Exclusion Criteria:

1. Subjects with a history of any illness, other than obesity, that may affect insulin sensitivity (anemia, infectious diseases, renal or hepatic failure, uncontrolled hypertension, cancer, lymphoma, chronic inflammatory conditions such as inflammatory bowel disease and rheumatoid arthritis, states of cortisol or growth hormone excess, alcoholism or drug abuse, and eating disorders).
2. History of diabetes mellitus.
3. Subjects taking any medications that are known to influence glucose metabolism such as glucocorticoids will also be excluded. We will screen for these conditions by means of a detailed history and review of systems and physical examination (see below).
4. Subjects taking any medications known to affect lipids such as statins will also be excluded. We will screen for these similar to above.
5. Cholesterol greater or equal to 250 mg/dL and/or triglyceride levels greater than 500 mg/dL at the time of screening, as determined by laboratory testing.
6. Subjects who have a known history of anaphylaxis or anaphylactoid-like reactions or who have a known hypersensitivity to anesthetic agents such as Lidocaine or Marcaine will be excluded from the study.
7. Hypersensitivity to fat emulsion or any component of the formulation; severe egg or legume (soybean) allergies; pathologic hyperlipidemia, lipoid nephrosis, acute pancreatitis associated with hyperlipemia.
8. Hypersensitivity to heparin or any component of the formulation
9. Severe thrombocytopenia, uncontrolled active bleeding, disseminated intravascular coagulation (DIC); suspected intracranial hemorrhage.
10. Subjects with a history of bleeding dyscrasia, poor wound healing or any medical condition precluding supine position will be excluded from the study.
11. Unable to follow study protocol or any condition that in the opinion of the investigator makes the subject unsuitable for the study.
12. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Changes of the plasma concentrations of Activins | 6 hours
  Area Under the Curve (AUC) of activins A, B, AB
Changes of the plasma concentrations of Follistatins | 6 hours
  Area Under the Curve (AUC) of follistatin, FSTL-3

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Kokkinos, MD, PhD, Principal Investigator — Medical School, National and Kapodistrian University of Athens, Laiko General Hospital
Locations (1):
- Diabetes Clinical Research Laboratory, 1st Department of Propaedeutic Internal Medicine, Athens, Greece

REFERENCES:
- [Derived] Perakakis N, Kokkinos A, Angelidi AM, Tsilingiris D, Gavrieli A, Yannakoulia M, Tentolouris N, Mantzoros CS. Circulating levels of five proglucagon-derived peptides in response to intravenous or oral glucose or lipids and to a mixed-meal in subjects with normal weight, overweight, and obesity. Clin Nutr. 2022 Sep;41(9):1969-1976. doi: 10.1016/j.clnu.2022.07.001. Epub 2022 Jul 19. PMID 35961260